CLINICAL TRIAL: NCT05223218
Title: Investigating the Diagnostic Potential of Tear Proteins in Breast, Ovarian, Prostate, Melanoma, Pancreatic, and Colon Cancer
Brief Title: Investigating the Diagnostic Potential of Tear Proteins in Cancer - A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Namida Lab (Industry)
Collaborators: Arkansas Urology (Unknown); CARTI (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB#56402
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer; Melanoma
Keywords: Preventative Screening; Protein Biomarkers; Lacrimal Tear Fluid; Non-invasive; Tear Collection; CLIA Laboratory; Affordable; Proteomics; Metabolomics; Protein Microarray; ELISA assay
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Lacrimal tear fluids will be stored for conducting pr
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Breast Cancer: Individuals aged between 18-100 years who are presenting for an evaluation of an abnormal exam or test (Mammogram, ultrasound, MRI, PET, etc.); presenting for the evaluation of a palpable lump or mass; presenting with a mass pre or post-biopsy as long as there is a portion of the mass remaining; or have been diagnosed with breast cancer but have not received treatment.
  Lacrimal tear fluid samples are collected using a Schirmer strip, a Class I Medical Device typically used to test for dry eye.
  Interventions: Other: Schirmer strip, a Class I Medical Device typically used to test for dry eye.
- Pancreatic Cancer: Individuals aged between 18-100 years who are presenting for an evaluation of an abnormal exam or test (Ultrasound, MRI, PET, etc.); presenting for the evaluation of a palpable lump or mass; presenting with a mass pre or post-biopsy as long as there is a portion of the mass remaining; or have been diagnosed with breast cancer but have not received treatment.
  Lacrimal tear fluid samples are collected using a Schirmer strip, a Class I Medical Device typically used to test for dry eye.
  Interventions: Other: Schirmer strip, a Class I Medical Device typically used to test for dry eye.
- Colon Cancer: Individuals aged between 18-100 years who are presenting for an evaluation of an abnormal exam or test (Ultrasound, MRI, PET, etc.); presenting for the evaluation of a palpable lump or mass; presenting with a mass pre or post-biopsy as long as there is a portion of the mass remaining; or have been diagnosed with breast cancer but have not received treatment.
  Lacrimal tear fluid samples are collected using a Schirmer strip, a Class I Medical Device typically used to test for dry eye.
  Interventions: Other: Schirmer strip, a Class I Medical Device typically used to test for dry eye.
- Prostate Cancer: Individuals aged between 18-100 years who are presenting for an evaluation of an abnormal exam or test (Ultrasound, MRI, PET, etc.); presenting for the evaluation of a palpable lump or mass; presenting with a mass pre or post-biopsy as long as there is a portion of the mass remaining; or have been diagnosed with breast cancer but have not received treatment.
  Lacrimal tear fluid samples are collected using a Schirmer strip, a Class I Medical Device typically used to test for dry eye.
  Interventions: Other: Schirmer strip, a Class I Medical Device typically used to test for dry eye.
- Melanoma: Individuals aged between 18-100 years who are presenting for an evaluation of an abnormal exam or test (Ultrasound, MRI, PET, etc.); presenting for the evaluation of a palpable lump or mass; presenting with a mass pre or post-biopsy as long as there is a portion of the mass remaining; or have been diagnosed with breast cancer but have not received treatment.
  Lacrimal tear fluid samples are collected using a Schirmer strip, a Class I Medical Device typically used to test for dry eye.
  Interventions: Other: Schirmer strip, a Class I Medical Device typically used to test for dry eye.
- Healthy Control: Individuals aged between 18-100 years who do not currently have a previous diagnosis of any cancer for which they are currently being treated.
  Lacrimal tear fluid samples are collected using a Schirmer strip, a Class I Medical Device typically used to test for dry eye.
  Interventions: Other: Schirmer strip, a Class I Medical Device typically used to test for dry eye.

INTERVENTIONS:
Other: Schirmer strip, a Class I Medical Device typically used to test for dry eye. — Schirmer strip is a Class I Medical Device typically used to test for dry eye and will be used to collect lacrimal tear fluids.

SUMMARY:
This Pilot Study is to investigate the tear proteins in a multitude of cancer types and indulge in biomarker discovery to manufacture simple, accurate, and novel tear-based diagnostic tests.

DETAILED DESCRIPTION:
The Pilot Study is an observational study to investigate the diagnostic potential of tear proteins for Breast, Ovarian, Prostate, Melanoma, Pancreatic, and Colon cancer. In this pilot study, we use lacrimal gland fluid (tears) as a liquid biopsy source for investigating the protein repertoire and conducting biomarker discovery studies with a goal to develop new tear-based tests that can detect crucial cancer-related biomarkers in the pan-cancer types.

Proteomic studies on tears have shown to express between 500-1500 proteins with ~35% overlap with serum proteome. The easy accessibility of tear fluid with minimal post-processing procedures and better access to lower molecular weight proteins make tears an ideal source to identify commonly associated cancer biomarkers.

Additionally, the results from this study will aid in improving our understanding of the cancer types and commonalities that exist between them.

ELIGIBILITY:
Inclusion Criteria:

* 18-100 years of age
* Presenting for the evaluation of an abnormal exam or test (mammogram, ultrasound, MRI, PET, etc.)
* Presenting for the evaluation of a palpable lump or mass
* Presenting with a mass may be pre or post-biopsy/diagnostic as long as there is a portion of the mass remaining.
* Have been diagnosed but have not received treatment

Exclusion Criteria:

* Less than 18 years of age OR more than 100 years of age
* Concurrent eye infection or trauma
* Acute conjunctivitis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population presented in the inclusion criteria will be recruited at multiple cancer centers and clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Identify Cancer-related Biomarkers | Dec 2023
  A tear protein repertoire will be created to identify key cancer biomarkers

SECONDARY OUTCOMES:
Tear Protein Concentrations | Dec 2023
  The total protein concentrations will be measured at different temperature conditions to determine the protein degradation profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Prashanth Ravishankar, PhD, Principal Investigator — Namida Lab Inc
Locations (1):
- Namida Lab, Fayetteville, Arkansas, United States